CLINICAL TRIAL: NCT05759520
Title: Phase III Clinical Trial to Evaluate the Immunogenicity and Safety of 13-valent Pneumococcal Conjugate Vaccine (Multivalent Conjugate) in Infants Aged 2 Months (at Least 6 Weeks) and 3 Months
Brief Title: Phase III Clinical Trial of 13-valent Pneumococcal Conjugate Vaccine (Multivalent Conjugate) in Infants
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fosun Adgenvax Biopharmaceutical Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ATG-PCV13-Ⅲ-2020001
Record Dates: First submitted 2023-02-26; First posted 2023-03-08 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Streptococcus Pneumoniae Infection
MeSH Terms: conditions — Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 2-month-old experimental group (Experimental): Vaccination of 4 doses of experimental vaccine(0,2,4,1 booster dose)
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine (multivalent conjugate)
- 2-month-old control group (Active Comparator): Vaccination of 4 doses of control vaccine(0,2,4,1 booster dose)
  Interventions: Biological: Prevenar 13
- 3-month-old group (Experimental): Vaccination of 4 doses of experimental vaccine(0,1,2,1 booster dose)
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine (multivalent conjugate)

INTERVENTIONS:
Biological: 13-valent pneumococcal conjugate vaccine (multivalent conjugate) — the 2-month-old experimental group and the 3-month-old group received the experimental vaccine
  Arms: 2-month-old experimental group; 3-month-old group
Biological: Prevenar 13 — the 2-month-old control group received the active control vaccine
  Arms: 2-month-old control group

SUMMARY:
This study is a phase III clinical trial to evaluate the immunogenicity and safety of the 13-valent pneumococcal conjugate vaccine (multivalent conjugate) in infants aged 2 months (at least 6 weeks) and 3 months. The main objectives of the study include: 1. To evaluate the immunogenicity of the trial vaccine in infants aged 2 months (at least 6 weeks) following the corresponding immunization schedule compared to the control vaccine; 2. To evaluate the immunogenicity of the trial vaccine in infants aged 3 months following the corresponding immunization schedule compared to the 2-month group; 3. To evaluate the safety of the trial vaccine in infants aged 2 months (at least 6 weeks) and 3 months following the corresponding immunization schedule.

ELIGIBILITY:
Inclusion Criteria:

Primary immunization phase:

1. The subject's legal guardian voluntarily agreed to allow his child to participate in the study and signed an informed consent form.
2. The subject's legal guardian has the ability to understand the study procedures and to participate in all planned follow-up visits.
3. Full-term pregnancy (37 weeks to 42 weeks gestation) and the birth weight was 2500g~4000g.
4. On the day of the first dose of vaccination, it meets the observation age of this clinical trial (2~3 months of age, with a minimum of 6 weeks) and be able to provide legal identification;
5. Not having received a non-live vaccine within 7 days prior to enrollment and not having received a live vaccine within 14 days;
6. The body temperature <37.5°C (axillary body temperature) on the day of enrollment.

Booster immunization phase:

1. Infants and children who have completed the full process of basic immunization in this clinical trial and are 12 to 15 months of age;
2. According to the opinion of the investigator, the subject's legal guardians and their families can comply with the requirements of the clinical trial protocol.

Exclusion Criteria:

Primary immunization phase:

1. The baby is born in abnormal labor (dystocia, instrumental delivery) or has a history of asphyxia and nervous system damage, and is now suffering from pathologic jaundice, perianal abscess and severe eczema;
2. Have been vaccinated against pneumococcus in the past or have a history of invasive diseases caused by pneumococcus in the past (confirmed by either clinical, serological or microbiological methods);
3. Previous history of severe allergy to any vaccine or drug, such as anaphylactic shock, allergic laryngeal edema, allergic purpura and local allergic necrosis reaction (Arthus reaction);
4. Suffering from congenital or acquired immunodeficiency, or receiving immunosuppressant treatment, such as systemic glucocorticoid treatment for more than 2 weeks one month before vaccination, such as prednisone or similar drugs > 5mg/day (use of local and inhaled/atomized steroids is eligible for enrollment);
5. Have received blood or blood-related products or immunoglobulin treatment before joining the group (hepatitis B immunoglobulin is acceptable);
6. Suffering from severe congenital malformation, severe developmental disorders, serious genetic diseases (such as severe thalassemia), severe malnutrition, etc.;
7. Suffering from infectious diseases such as tuberculosis and viral hepatitis, or parents infected with human immunodeficiency virus;
8. Having contraindications to intramuscular injections such as thrombocytopenia, any coagulation disorder or receiving anticoagulant therapy;
9. Those with a history or family history of convulsions, epilepsy, encephalopathy and psychosis;
10. Asplenia, functional asplenia, and asplenia or splenectomy for any reason;
11. Subjects with other safety risks or conditions that, in the opinion of the investigator, may interfere with the assessment of the purpose of the study.

Booster immunization phase:

1. Subject received any other pneumonia vaccine after primary immunization and before booster immunization;
2. Subject has received blood or blood-related products or immunoglobulin treatment within 3 months before booster immunization;
3. The subjects have known or suspected immunological functional defects since they participated in this clinical trial, including receiving immunosuppressant treatment (such as systemic glucocorticoid treatment for more than 2 weeks in one month before vaccination, such as prednisone or similar drugs > 5mg/day) and their parents are HIV-infected;
4. According to the researcher's judgment, the subjects have any other factors that are not suitable for clinical trials.

Ages: 6 Weeks to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1800 (Estimated)
Dates: Start 2022-11-04 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
seroprotection rate of 13 vaccine serotype-specific pneumococcal IgG antibodies | 30 days after primary immunization
  Immunogenicity
13 vaccine serotype-specific pneumococcal IgG antibodies GMC | 30 days after primary immunization
  Immunogenicity
incidence of adverse events (AE) | 30 minutes/0~7 days/0~30 days after each dose of vaccination
  Safety
incidence of all serious adverse events (SAEs) | from the first dose to 6 months after primary immunization
  Safety
incidence of all serious adverse events (SAEs) | from the first dose of vaccination to 12 months after the booster immunization
  Safety

SECONDARY OUTCOMES:
percentage of subjects with 13 vaccine serotype-specific pneumococcal IgG antibody concentrations ≥1.0 μg/ml | 30 days after primary immunization
  Primary stage
the positivity rate of pneumococcal OPA antibodies for 13 vaccine serotypes | 30 days after primary immunization
  Primary stage
the GMT of pneumococcal OPA antibodies for 13 vaccine serotypes | 30 days after primary immunization
  Primary stage
the seroconversion rate of pneumococcal OPA antibodies for 13 vaccine serotypes | 30 days after primary immunization
  Primary stage
seroprotection rate of 13 vaccine serotype-specific pneumococcal IgG antibodies | 30 days after booster immunization
  Booster stage
percentage of subjects with 13 vaccine serotype-specific pneumococcal IgG antibody concentrations ≥ 1.0 μg/mL | 30 days after booster immunization
  Booster stage
GMC of 13 vaccine serotype-specific pneumococcal IgG antibodies | 30 days after booster immunization
  Booster stage
the positivity rate of pneumococcal OPA antibodies for 13 vaccine serotypes | 30 days after booster immunization
  Booster stage
the GMT of pneumococcal OPA antibodies for 13 vaccine serotypes | 30 days after booster immunization
  Booster stage

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Yizhou District Disease Prevention Control Center, Hechi, Guangxi
  - Zhongshan County Center for Disease Control and Prevention, Hezhou, Guangxi
  - Luzhai County Disease Prevention Control Center, Liuchow, Guangxi
  - Binyang County Center for Disease Control and Prevention, Nanning, Guangxi
  - Wuming District Center for Disease Control and Prevention, Nanning, Guangxi

IPD SHARING:
Plan to Share IPD: No